CLINICAL TRIAL: NCT03970018
Title: ADPKD Patients and Peritoneal Dialysis: Creation and Validation of Predictive Score for Peritoneal Pressure
Brief Title: ADPKD and Peritoneal Dialysis: How Anticipate Peritoneal Pressure?
Acronym: PDP-ADPKD
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PA18042
Record Dates: First submitted 2018-03-27; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Autosomal dominant polycystic kidney disease; peritoneal dialysis; peritoneal pressure
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Autosomal dominant polycystic kidney disease: Autosomal dominant polycystic kidney disease (ADPKD) patients starting peritoneal dialysis for end stage renal failure will be included in this study.
  Interventions: Other: Intra-peritoneal pressure

INTERVENTIONS:
Other: Intra-peritoneal pressure — Measurement of intra-peritoneal pressure

SUMMARY:
Autosomal dominant polycystic kidney disease (ADPKD) is first genetic kidney disease and fourth etiology of end stage renal disease in the world. Peritoneal dialysis is underuse in this population. Indeed in this pathology, behind big kidneys and big liver, a hyper pressure is feared with technical failure. The lack of abdominal space could generate increase of peritoneal pressure. Hyper pressure is already known to be a risk factor of technical failure and over mortality in peritoneal dialysis patients (all nephropathies included). It depends on body mass index and body surface modulating injected volume for each patient. Anticipate peritoneal pressure in this population ADPKD could be an important information for distinguish those who can use peritoneal dialysis without fear and those at risk of technical failure.

The primary objective is to create and validate prediction score for intra-peritoneal pressure, in peritoneal dialysis for ADPKD patients thanks to clinical and radiological values.

The secondary objectives are to study the association between intra-peritoneal pressure and patient's outcome (global survival and technical survival).

Retrospective, multicentric, national, cohort study will be performed. For the first step (score creation): ADPKD patients starting peritoneal dialysis for end stage renal failure between 01/01/2010 and 31/12/2015 with tomodensitometry between one year before beginning and one year after were included.

For the second step (score validation): ADPKD patients starting peritoneal dialysis for end stage renal failure between 01/01/2016 and 31/12/2017 with tomodensitometry between one year before beginning and one year after were included.

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease (ADPKD) is first genetic kidney disease and fourth etiology of end stage renal disease in the world. Peritoneal dialysis is underuse in this population. Indeed in this pathology, behind big kidneys and big liver, a hyper pressure is feared with technical failure. The lack of abdominal space could generate increase of peritoneal pressure. Hyper pressure is already known to be a risk factor of technical failure and over mortality in peritoneal dialysis patients (all nephropathies included). It depends on body mass index and body surface modulating injected volume for each patient. Anticipate peritoneal pressure in this population ADPKD could be an important information for distinguish those who can use peritoneal dialysis without fear and those at risk of technical failure.

The primary objective is to create and validate prediction score for intra-peritoneal pressure, in peritoneal dialysis for ADPKD patients thanks to clinical and radiological values.

The secondary objectives are to study the association between intra-peritoneal pressure and patient's outcome (global survival and technical survival).

Retrospective, multicentric, national, cohort study will be performed. For the first step (score creation): ADPKD patients starting peritoneal dialysis for end stage renal failure between 01/01/2010 and 31/12/2015 with tomodensitometry between one year before beginning and one year after will be included.

For the second step (score validation): ADPKD patients starting peritoneal dialysis for end stage renal failure between 01/01/2016 and 31/12/2017 with tomodensitometry between one year before beginning and one year after will be included.

Data regarding organ volume and clinical data wich can influence pressure and patient's outcome (global survival and technical survival) will be recorded.

A bivariate analysis will be performed to study the association between intra-peritoneal pressure and clinical data. A multivariate analysis by multiple linear regressions will be performed to create the score. Survival analysis by log rank test and cox regression model will be performed for global survival and technical survival.

ELIGIBILITY:
Inclusion criteria:

* Major ADPKD patients starting peritoneal dialysis for end stage renal disease between 2010 January 1st and 2015 December 31
* Must have an abdominal tomodensitometry in 2 years around start (between 1 year before and 1 year after)
* Must have an intraperitoneal pressure measurement in the first year of peritoneal dialysis.
* Major ADPKD patients starting peritoneal dialysis for end stage renal disease between 2015 January 1st and 2017 December 31

Non-inclusion criteria:

* Lack of tomodensitometry or intraperitoneal pressure.
* History of nephrectomy or arterioembolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Autosomal dominant polycystic kidney disease (ADPKD) patients starting peritoneal dialysis for end stage renal failure
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Creation of a predictive score of intra-peritoneal pressure | Day 0
  Data regarding organ volume and clinical data wich can influence intra-peritoneal pressure will be recorded. A bivariate analysis will be performed to study the association between intra-peritoneal pressure and clinical data. A multivariate analysis by multiple linear regressions will be performed.
Validation of a predictive score of intraperitoneal pressure | Day 0
  Measurment and calculation of intraperitoneal pressure

SECONDARY OUTCOMES:
Global survival | 12 months
  Data regarding global survival will be recorded 12 months after the beginning of peritoneal dialysis.
Technical survival | 12 months
  Data regarding technical survival will be recorded 12 months after the beginning of peritoneal dialysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France